CLINICAL TRIAL: NCT02761629
Title: Randomized, Multi-Center, Phase IV, Comparative Study to Assess the Efficacy and Safety of Combined Peg-Interferon Alpha-2a (40 kD) With Ribavirin Combined Therapy for 48 or 72 Weeks of Treatment and 24 Weeks of Follow-Up in Patients With Chronic Hepatitis C, Genotype 1, Co-Infected With Human Immunodeficiency Virus
Brief Title: Efficacy and Safety of Peg-Interferon Alpha-2a Plus Ribavirin in Genotype 1 Chronic Hepatitis C Participants Co-Infected With Human Immunodeficiency Virus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML18473
Record Dates: First submitted 2016-05-03; First posted 2016-05-04 (Estimated); Results first posted 2016-08-16 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-07

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

ARMS (2):
- Peg-IFN-Alpha-2A+Ribavirin - 48 Weeks (Experimental): Participants will receive Peg-IFN-Alpha-2A and ribavirin for 48 weeks.
  Interventions: Drug: Peg-Interferon Alpha-2A; Drug: Ribavirin
- Peg-IFN-Alpha-2A+Ribavirin - 72 Weeks (Active Comparator): Participants will receive Peg-IFN-Alpha-2A and ribavirin for 72 weeks.
  Interventions: Drug: Peg-Interferon Alpha-2A; Drug: Ribavirin

INTERVENTIONS:
Drug: Peg-Interferon Alpha-2A — Peg-IFN-Alpha-2A will be administered at 180 micrograms (mcg) once weekly via subcutaneous injection.
  Other Names: Pegasys, Peg-IFN-Alpha-2A
Drug: Ribavirin — Ribavirin will be administered as either 1000 milligrams (mg) (2*200 mg tablets in morning and 3*200 mg tablets in evening) for participants weighing less than (<) 75 kilograms (kg) or as 1200 mg (3*200 mg tablets in morning and 3*200 mg tablets in evening) for participants weighing greater than or equal to (>/=) 75 kg.

SUMMARY:
This randomized, multi-center, Phase IV, comparative study will assess the efficacy and safety of combined peg-interferon alpha-2a (Peg-IFN-Alpha-2A) and ribavirin therapy for 48 or 72 weeks of treatment and 24 weeks of follow-up in participants with Genotype 1 chronic hepatitis C (CHC), co-infected with human immunodeficiency virus type 1 (HIV-1).

ELIGIBILITY:
Inclusion Criteria:

* Serological evidence of chronic hepatitis C infection by anti-hepatitis C virus (HCV) test
* Detectable HCV-ribonucleic acid (RNA) plasma level testing by Roche AMPLICOR HCV (<50 International Units per milliliter [IU/mL]) (qualitative test)
* Chronic liver disease consistent with infection of CHC
* Compensated liver disease (Child-Pugh Grade A)
* Serological evidence of infection by HIV-1 test, anti-HIV-1 or HIV-1 RNA detection
* Negative pregnancy urine or blood test (for women in childbearing age); additionally, all men and women of childbearing potential must agree to use two effective forms of contraception during the treatment and during the 6 months after the end of treatment

Exclusion Criteria:

* Pregnant or nursing women and male partners of pregnant women
* Prior therapy with interferon (IFN) or ribavirin and any investigational medication less than or equal to (</=) 6 weeks before the first dose of the study drug
* History or other evidence of a medical condition associated with chronic liver disease further than HCV
* Active opportunistic infection associated with HIV and / or cancer requiring systemic therapy
* History of any other significant illness which in the investigator's opinion, could result in the participant's inability to meet the Protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2005-04; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (12):
- Brazil (12):
  - Campinas
  - Florianópolis
  - Itajaí
  - Juiz de Fora
  - Porto Alegre
  - Recife
  - Ribeirão Preto
  - Rio de Janeiro
  - Rio Grande
  - Santo André
  - Santos
  - São Paulo

RESULTS

PARTICIPANT FLOW:
Groups:
- Peg-IFN-Alpha-2A+Ribavirin - 48 Weeks: Participants received peg-interferon alpha-2A (Peg-IFN-Alpha-2A) and ribavirin for 48 weeks. Peg-IFN-Alpha-2A was administered at 180 micrograms (mcg) once weekly via subcutaneous injection. Ribavirin was administered as either 1000 milligrams (mg) per day (2*200 mg tablets in morning and 3*200 mg tablets in evening) for participants weighing less than (<) 75 kilograms (kg) or as 1200 mg per day (3*200 mg tablets in morning and 3*200 mg tablets in evening) for participants weighing greater than or equal to (>/=) 75 kg.
- Peg-IFN-Alpha-2A+Ribavirin - 72 Weeks: Participants received Peg-IFN-Alpha-2A and ribavirin for 72 weeks. Peg-IFN-Alpha-2A was administered at 180 mcg once weekly via subcutaneous injection. Ribavirin was administered as either 1000 mg per day (2*200 mg tablets in morning and 3*200 mg tablets in evening) for participants weighing <75 kg or as 1200 mg per day (3*200 mg tablets in morning and 3*200 mg tablets in evening) for participants weighing >/=75 kg.
Period: Overall Study
Arm/Group | Peg-IFN-Alpha-2A+Ribavirin - 48 Weeks | Peg-IFN-Alpha-2A+Ribavirin - 72 Weeks
Started | 90 | 90
Treated | 82 | 86
Completed | 63 | 58
Not Completed | 27 | 32
Not completed — Adverse Event/Intercurrent Illness | 7 | 5
Not completed — Insufficient Therapeutic Response | 2 | 7
Not completed — Failure to Return | 2 | 4
Not completed — Did not Cooperate/Refused Treatment | 2 | 4
Not completed — Protocol Violation | 2 | 2
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Other | 0 | 2
Not completed — Lost to Follow-up | 4 | 1
Not completed — Randomized But Not Treated | 8 | 4

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis population included all randomized participants who receive at least one dose of any study medication and have at least one post-baseline efficacy assessment.
Groups:
- Peg-IFN-Alpha-2A+Ribavirin - 48 Weeks: Participants received Peg-IFN-Alpha-2A and ribavirin for 48 weeks. Peg-IFN-Alpha-2A was administered at 180 mcg once weekly via subcutaneous injection. Ribavirin was administered as either 1000 mg per day (2*200 mg tablets in morning and 3*200 mg tablets in evening) for participants weighing <75 kilograms (kg) or as 1200 mg per day (3*200 mg tablets in morning and 3*200 mg tablets in evening) for participants weighing >/=75 kg.
- Total: Total of all reporting groups
Arm/Group | Peg-IFN-Alpha-2A+Ribavirin - 48 Weeks | Peg-IFN-Alpha-2A+Ribavirin - 72 Weeks | Total
Number analyzed (Participants) | 80 | 85 | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (7.9) | 42.2 (8.4) | 42.3 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 26 | 57
  Male | 49 | 59 | 108

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR)
Description: SVR was defined as having un-detectable hepatitis C virus (HCV) ribonucleic acid (RNA) levels 24 weeks after completion of study treatment. HCV RNA levels were measured using Roche COBAS AMPLICOR HCV Test (limit of detection: 50 International Units per milliliter [IU/mL]). Participants with detectable HCV RNA or without measurement at the end of the 24 week after completion of study treatment were considered as non-responders.
Time Frame: 24 weeks after completion of study treatment (up to Week 72 for "Peg-IFN-Alpha-2A+Ribavirin - 48 Weeks" arm and up to Week 96 for "Peg-IFN-Alpha-2A+Ribavirin - 72 Weeks" arm)
Population: Intent-to-treat (ITT) analysis population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Peg-IFN-Alpha-2A+Ribavirin - 48 Weeks | Peg-IFN-Alpha-2A+Ribavirin - 72 Weeks
Number analyzed (Participants) | 80 | 85
percentage of participants | 23.8 [15.0 to 34.6] | 36.5 [26.3 to 47.6]
Statistical Analysis 1: Comparison: Peg-IFN-Alpha-2A+Ribavirin - 48 Weeks vs Peg-IFN-Alpha-2A+Ribavirin - 72 Weeks; Test type: Superiority or Other; p = 0.0536, Fisher Exact; Difference in Response Rates = 12.7, 95% CI 2-sided [-0.01 to 26.6] — Exact 95% confidence interval was from the binomial distribution for response rate

2. Secondary Outcome: Percentage of Participants With Undetectable HCV RNA
Description: HCV RNA levels were measured using Roche COBAS AMPLICOR HCV Test (limit of detection: 50 IU/mL). Data for this outcome measure was to be reported up to end of treatment visit (Week 48 for 'Peg-IFN-Alpha-2A+Ribavirin - 48 Weeks' arm and Week 72 for 'Peg-IFN-Alpha-2A+Ribavirin - 72 Weeks' arm).
Time Frame: For "Peg-IFN-Alpha-2A+Ribavirin - 48 Weeks" arm: Weeks 4, 12, 24, and 48; for "Peg-IFN-Alpha-2A+Ribavirin - 72 Weeks" arm: Weeks 4, 12, 24, 48, and 72
Population: ITT analysis population. Here, number of participants analyzed = participants who were evaluable for this outcome and "n" = participants who were evaluable for this outcome at specified time-point; for each arm, respectively.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Peg-IFN-Alpha-2A+Ribavirin - 48 Weeks | Peg-IFN-Alpha-2A+Ribavirin - 72 Weeks
Number analyzed (Participants) | 73 | 83
percentage of participants
  Week 4 (n=73, 83) | 2.7 [0.3 to 9.6] | 12.0 [5.9 to 21.0]
  Week 12 (n=73, 81) | 23.3 [14.2 to 34.7] | 28.4 [18.9 to 39.5]
  Week 24 (n=73, 78) | 52.1 [40.0 to 63.9] | 53.8 [42.2 to 65.2]
  Week 48 (n=68, 71) | 55.9 [43.3 to 67.9] | 64.8 [52.5 to 75.8]
  Week 72 (n=0, 65) | NA [NA to NA] — Data for this outcome measure was to be reported up to end of treatment visit (Week 48 for this arm); hence, no data reported for Week 72 for this arm. | 56.9 [44.0 to 69.2]

3. Secondary Outcome: Percentage of Participants With Undetectable HCV RNA 12 Weeks After the Last Dose of Peg-IFN-Alpha-2A
Description: HCV RNA levels were measured using Roche COBAS AMPLICOR HCV Test (limit of detection: 50 IU/mL). Participants with detectable HCV RNA or without measurement at the end of 12 weeks after the last dose of Peg-IFN-Alpha-2A were considered as non-responders.
Time Frame: 12 weeks after the last dose of Peg-IFN-Alpha-2A (up to Week 60 for "Peg-IFN-Alpha-2A+Ribavirin - 48 Weeks" arm and up to Week 84 for "Peg-IFN-Alpha-2A+Ribavirin - 72 Weeks" arm)
Population: ITT analysis population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Peg-IFN-Alpha-2A+Ribavirin - 48 Weeks | Peg-IFN-Alpha-2A+Ribavirin - 72 Weeks
Number analyzed (Participants) | 80 | 85
percentage of participants | 23.8 [15.0 to 34.6] | 36.5 [26.3 to 47.6]

4. Secondary Outcome: Percentage of Participants Without SVR Among Participants With Undetectable HCV RNA at the End of Treatment
Description: SVR was defined as having undetectable HCV RNA levels 24 weeks after completion of study treatment. HCV RNA levels were measured using Roche COBAS AMPLICOR HCV Test (limit of detection: 50 IU/mL). Percentage of participants without SVR among participants with undetectable HCV RNA at the end of treatment was reported (end of treatment = Week 48 for "Peg-IFN-Alpha-2A+Ribavirin - 48 Weeks" arm and Week 72 for "Peg-IFN-Alpha-2A+Ribavirin - 72 Weeks" arm).
Time Frame: as for outcome 1
Population: ITT analysis population. Here, number of participants analyzed signifies participants with undetectable HCV RNA at the end of treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Peg-IFN-Alpha-2A+Ribavirin - 48 Weeks | Peg-IFN-Alpha-2A+Ribavirin - 72 Weeks
Number analyzed (Participants) | 38 | 37
percentage of participants | 52.6 | 24.3
Statistical Analysis 1: Comparison: Peg-IFN-Alpha-2A+Ribavirin - 48 Weeks vs Peg-IFN-Alpha-2A+Ribavirin - 72 Weeks; Test type: Superiority or Other; p = 0.0175, Fisher Exact

5. Secondary Outcome: Serum Human Immunodeficiency Virus (HIV) RNA Levels
Description: HIV RNA levels were measured using Roche AMPLICOR MONITOR HIV-1 Test (limit of detection: 400 HIV-1 RNA copies/mL). Data for this outcome measure was to be reported up to 24 weeks after end of treatment visit (Week 72 for 'Peg-IFN-Alpha-2A+Ribavirin - 48 Weeks' arm and Week 96 for 'Peg-IFN-Alpha-2A+Ribavirin - 72 Weeks' arm).
Time Frame: For "Peg-IFN-Alpha-2A+Ribavirin - 48 Weeks" arm: Weeks 4, 12, 24, 48, and 72; for "Peg-IFN-Alpha-2A+Ribavirin - 72 Weeks" arm: Weeks 4, 12, 24, 48, 72, and 96
Population: ITT analysis population. Here, number of participants analyzed = participants with detectable HIV RNA levels and "n" = participants with detectable HIV RNA levels at specified time-point; for each arm, respectively.
Measure: Mean (Standard Deviation); unit: Log10 copies per milliliter
Arm/Group | Peg-IFN-Alpha-2A+Ribavirin - 48 Weeks | Peg-IFN-Alpha-2A+Ribavirin - 72 Weeks
Number analyzed (Participants) | 12 | 23
Log10 copies per milliliter
  Baseline (n=12, 23) | 4.23 (0.82) | 4.64 (0.74)
  Week 4 (n=6, 16) | 3.94 (0.38) | 3.98 (0.69)
  Week 24 (n=9, 20) | 3.96 (0.36) | 4.21 (0.72)
  Week 48 (n=11, 17) | 4.02 (0.65) | 4.41 (0.75)
  Week 72 (n=10, 9) | 4.08 (0.78) | 4.51 (0.85)
  Week 96 (n=0, 13) | NA (NA) — Data for this outcome measure was to be reported up to 24 weeks after end of treatment (Week 72 for this arm); hence, no data reported for Week 96 for this arm. | 4.22 (0.85)

6. Secondary Outcome: Change From Baseline in Cluster of Differentiation (CD) 4 (CD4) Cell Counts at Weeks 4, 12, 24, 48, 72, and 96
Description: Data for this outcome measure was to be reported up to 24 weeks after end of treatment visit (Week 72 for 'Peg-IFN-Alpha-2A+Ribavirin - 48 Weeks' arm and Week 96 for 'Peg-IFN-Alpha-2A+Ribavirin - 72 Weeks' arm).
Time Frame: For "Peg-IFN-Alpha-2A+Ribavirin - 48 Weeks" arm: Baseline, Weeks 4, 12, 24, 48, and 72; for "Peg-IFN-Alpha-2A+Ribavirin - 72 Weeks" arm: Baseline, Weeks 4, 12, 24, 48, 72, and 96
Population: ITT analysis population. Here, number of participants analyzed = participants who were evaluable for this outcome and "n" = participants who were evaluable at specified time-point; for each arm, respectively.
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter (cells/mm^3)
Arm/Group | Peg-IFN-Alpha-2A+Ribavirin - 48 Weeks | Peg-IFN-Alpha-2A+Ribavirin - 72 Weeks
Number analyzed (Participants) | 78 | 81
Cells per cubic millimeter (cells/mm^3)
  Baseline (n=78, 81) | 578.7 (277.1) | 546.2 (278.8)
  Change at Week 4 (n=69, 74) | -148.2 (197.5) | -88.0 (154.9)
  Change at Week 12 (n=68, 75) | -185.4 (192.7) | -164.5 (193.9)
  Change at Week 24 (n=69, 68) | -206.7 (217.0) | -178.4 (207.5)
  Change at Week 48 (n=61, 67) | -209.4 (242.4) | -196.4 (226.4)
  Change at Week 72 (n=58, 55) | 9.5 (188.9) | -167.5 (235.8)
  Change at Week 96 (n=0, 62) | NA (NA) — Data for this outcome measure was to be reported up to 24 weeks after end of treatment (Week 72 for this arm); hence, no data reported for Week 96 for this arm. | -15.1 (212.2)

7. Secondary Outcome: Change From Baseline in CD4/CD8 Ratio at Weeks 4, 12, 24, 48, 72, and 96
Description: as for outcome 6
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Peg-IFN-Alpha-2A+Ribavirin - 48 Weeks | Peg-IFN-Alpha-2A+Ribavirin - 72 Weeks
Number analyzed (Participants) | 78 | 81
Ratio
  Baseline (n=78, 81) | 0.67 (0.39) | 0.68 (0.44)
  Change at Week 4 (n=69, 74) | 0.11 (0.42) | 0.09 (0.21)
  Change at Week 12 (n=68, 75) | 0.22 (0.31) | 0.20 (0.27)
  Change at Week 24 (n=69, 68) | 0.36 (0.51) | 0.29 (0.30)
  Change at Week 48 (n=61, 67) | 0.43 (0.47) | 0.30 (0.43)
  Change at Week 72 (n=58, 55) | 0.12 (0.41) | 0.36 (0.43)
  Change at Week 96 (n=0, 62) | NA (NA) — Data for this outcome measure was to be reported up to 24 weeks after end of treatment (Week 72 for this arm); hence, no data reported for Week 96 for this arm. | 0.09 (0.35)

8. Secondary Outcome: Percentage of Participants With Alanine Aminotransferase (ALT) Level Categories
Description: ALT levels were classified as: Normal Limit (NL) (as per laboratory standard), >1-2 Upper Normal Limit (ULN), >2-5 ULN, >5-10 ULN, and >10 ULN. Percentage of participants in each of these ALT level categories was reported. Data for this outcome measure was to be reported up to 24 weeks after end of treatment visit (Week 72 for 'Peg-IFN-Alpha-2A+Ribavirin - 48 Weeks' arm and Week 96 for 'Peg-IFN-Alpha-2A+Ribavirin - 72 Weeks' arm).
Time Frame: as for outcome 5
Population: Safety analysis population: all randomized participants who receive >/=1 dose of any study medication and had >/=1 post-baseline safety assessment. Number of participants analyzed= overall participants who were evaluable for this outcome at any time-point and "n" = participants who were evaluable at specified time-point; for each arm, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Peg-IFN-Alpha-2A+Ribavirin - 48 Weeks | Peg-IFN-Alpha-2A+Ribavirin - 72 Weeks
Number analyzed (Participants) | 79 | 82
percentage of participants
  Week 4, NL (n=70, 78) | 50.0 | 52.6
  Week 4, >1-2 ULN (n=70, 78) | 40.0 | 38.5
  Week 4, >2-5 ULN (n=70, 78) | 10.0 | 9.0
  Week 4, >5-10 ULN (n=70, 78) | 0.0 | 0.0
  Week 4, >10 ULN (n=70, 78) | 0.0 | 0.0
  Week 12, NL (n=76, 77) | 61.8 | 62.3
  Week 12, >1-2 ULN (n=76, 77) | 27.6 | 29.9
  Week 12, >2-5 ULN (n=76, 77) | 10.5 | 5.2
  Week 12, >5-10 ULN (n=76, 77) | 0.0 | 1.3
  Week 12, >10 ULN (n=76, 77) | 0.0 | 1.3
  Week 24, NL (n=74, 74) | 70.3 | 63.5
  Week 24, >1-2 ULN (n=74, 74) | 27.0 | 28.4
  Week 24, >2-5 ULN (n=74, 74) | 2.7 | 6.8
  Week 24, >5-10 ULN (n=74, 74) | 0.0 | 0.0
  Week 24, >10 ULN (n=74, 74) | 0.0 | 1.4
  Week 48, NL (n=65, 71) | 67.7 | 69.0
  Week 48, >1-2 ULN (n=65, 71) | 24.6 | 26.8
  Week 48, >2-5 ULN (n=65, 71) | 7.7 | 2.8
  Week 48, >5-10 ULN (n=65, 71) | 0.0 | 1.4
  Week 48, >10 ULN (n=65, 71) | 0.0 | 0.0
  Week 72, NL (n=59, 61) | 52.5 | 68.9
  Week 72, >1-2 ULN (n=59, 61) | 27.1 | 27.9
  Week 72, >2-5 ULN (n=59, 61) | 20.3 | 3.3
  Week 72, >5-10 ULN (n=59, 61) | 0.0 | 0.0
  Week 72, >10 ULN (n=59, 61) | 0.0 | 0.0
  Week 96, NL (n=0, 62) | NA — Data for this outcome measure was to be reported up to 24 weeks after end of treatment (Week 72 for this arm); hence, no data reported for Week 96 for this arm. | 50.0
  Week 96, >1-2 ULN (n=0, 62) | NA — Data for this outcome measure was to be reported up to 24 weeks after end of treatment (Week 72 for this arm); hence, no data reported for Week 96 for this arm. | 35.5
  Week 96, >2-5 ULN (n=0, 62) | NA — Data for this outcome measure was to be reported up to 24 weeks after end of treatment (Week 72 for this arm); hence, no data reported for Week 96 for this arm. | 12.9
  Week 96, >5-10 ULN (n=0, 62) | NA — Data for this outcome measure was to be reported up to 24 weeks after end of treatment (Week 72 for this arm); hence, no data reported for Week 96 for this arm. | 1.6
  Week 96, >10 ULN (n=0, 62) | NA — Data for this outcome measure was to be reported up to 24 weeks after end of treatment (Week 72 for this arm); hence, no data reported for Week 96 for this arm. | 0.0

ADVERSE EVENTS:
Time Frame: 96 weeks
Description: Safety analysis population.
Arm/Group | Peg-IFN-Alpha-2A+Ribavirin - 48 Weeks | Peg-IFN-Alpha-2A+Ribavirin - 72 Weeks
Serious Adverse Events (participants affected / at risk) | 7/82 | 12/86
Other Adverse Events (participants affected / at risk) | 79/82 | 81/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peg-IFN-Alpha-2A+Ribavirin - 48 Weeks (N=82) | Peg-IFN-Alpha-2A+Ribavirin - 72 Weeks (N=86)
Pneumonia NOS (Infections and infestations) | 1 | 0
Postoperative infection (Infections and infestations) | 1 | 0
Respiratory tract infection NOS (Infections and infestations) | 1 | 1
Cytomegalovirus oesophagitis (Infections and infestations) | 0 | 1
Furuncle (Infections and infestations) | 0 | 1
Mycobacterial infection NOS (Infections and infestations) | 0 | 1
Diarrhoea NOS (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Lip and/or oral cavity cancer NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pregnancy NOS (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Irritability (Psychiatric disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Anaemia not otherwise specified (NOS) (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Erythema of eyelid (Eye disorders) | 0 | 1
Cholecystitis NOS (Hepatobiliary disorders) | 0 | 1
Hepatic disorder NOS (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Vulvar dysplasia (Reproductive system and breast disorders) | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1
Drug abuser NOS (Social circumstances) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Peg-IFN-Alpha-2A+Ribavirin - 48 Weeks (N=82) | Peg-IFN-Alpha-2A+Ribavirin - 72 Weeks (N=86)
Anaemia NOS (Blood and lymphatic system disorders) | 31 | 25
Neutropenia (Blood and lymphatic system disorders) | 13 | 14
Nausea (Gastrointestinal disorders) | 21 | 20
Diarrhoea NOS (Gastrointestinal disorders) | 13 | 16
Abdominal pain upper (Gastrointestinal disorders) | 10 | 8
Vomiting NOS (Gastrointestinal disorders) | 9 | 17
Dyspepsia (Gastrointestinal disorders) | 5 | 7
Abdominal pain NOS (Gastrointestinal disorders) | 4 | 9
Pyrexia (General disorders) | 30 | 32
Fatigue (General disorders) | 26 | 27
Asthenia (General disorders) | 23 | 30
Influenza like illness (General disorders) | 13 | 12
Malaise (General disorders) | 10 | 8
Chest pain (General disorders) | 8 | 6
Influenza (Infections and infestations) | 6 | 7
Sinusitis NOS (Infections and infestations) | 6 | 7
Herpes simplex (Infections and infestations) | 5 | 3
Oral candidiasis (Infections and infestations) | 4 | 5
Weight decreased (Investigations) | 9 | 8
Anorexia (Metabolism and nutrition disorders) | 25 | 22
Appetite decreased NOS (Metabolism and nutrition disorders) | 9 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 38 | 33
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 9
Headache (Nervous system disorders) | 34 | 41
Dizziness (Nervous system disorders) | 14 | 8
Somnolence (Nervous system disorders) | 6 | 8
Depression (Psychiatric disorders) | 16 | 11
Irritability (Psychiatric disorders) | 15 | 13
Insomnia (Psychiatric disorders) | 14 | 23
Anxiety (Psychiatric disorders) | 8 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 11
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.